CLINICAL TRIAL: NCT02085629
Title: The ONE Study: A Unified Approach to Evaluating Cellular Immunotherapy in Solid Organ Transplantation - M Reg Trial
Brief Title: The ONE Study M Reg Trial
Acronym: ONEmreg12
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Insufficient rate of patient recruitment and treatment.
Sponsor: University of Regensburg (Other)
Responsible Party: Principal Investigator, Edward Geissler, Professor, University of Regensburg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONEmreg12; 2013-000999-15 (EudraCT Number); grant number 260687 (Other Grant/Funding Number: European Union FP7 Programme)
Record Dates: First submitted 2014-03-10; First posted 2014-03-13 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Renal Failure, End Stage
Keywords: renal failure, end stage; renal transplantation; cell therapy; macrophages, monocyte derived; immune tolerance; ONE Study; immunotherapy
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- M reg treatment (Experimental): Donor M reg (2.5-7.5 million cells/kg) IV infused (6-7d before Tx) into recipients of a LD renal Tx. Recipients also receive prednisolone, mycophenolate mofetil and tacrolimus, as detailed below:
  Prednisolone
  * D 0: 500 mg IV
  * D 1: 125 mg IV
  * D 2 - 14: 20.0 mg/d (oral)
  * Wk 3 - 4: 15.0 mg/d
  * Wk 5 - 8: 10.0 mg/d
  * Wk 9 - 12: 5.0 mg/d
  * Wk 13 - 14: 2.5 mg/d
  * Wk 15 - End: Cessation
  MMF (or biologic equiv.)
  * D -7 to -2: 500 mg/d (250mg 2x/d)
  * D -1 to 14: 2000 mg/d
  * Wk 3 - 36: 1000 mg/d
  * Wk 37 - 40: 750 mg/d
  * Wk 41 - 44: 500 mg/d
  * Wk 45 - 48: 250 mg/d
  * Wk 49 - End: Cessation NOTE: MMF tapering will only happen if a 36-Wk biopsy shows no signs of subclinical rejection or if there is no evidence of declining renal function or if the clinician has any other concern about dose reduction.
  Tacrolimus (or biologic equiv.)
  * ≤ 48 h pre-Tx to D 14: 3-12 ng/ml
  * Wk 3 - 12: 3-10 ng/ml
  * Wk 13 - 36: 3-8 ng/ml
  * Wk 37 - End: 3-6 ng/ml
  Interventions: Biological: Donor M reg (Mreg_UKR)

INTERVENTIONS:
Biological: Donor M reg (Mreg_UKR) — Experimental: M reg treatment
  Donor M reg (2.5-7.5 million cells/kg) IV infused (6-7d before Tx) into recipients of a living donor renal Tx. Recipients also receive prednisolone, mycophenolate mofetil and tacrolimus background immunosuppression (as described in detail in the arm description).

SUMMARY:
To collect evidence of the safety of administering donor-derived regulatory macrophage (M reg) preparations to living-donor renal transplant recipients in the context of an international European Union funded consortium aimed at evaluating cellular immunotherapy in solid organ transplantation (The ONE Study). It is anticipated that immune regulation induced by M reg therapy can eventually be used to reduce the need for conventional immunosuppression in transplant recipients.

DETAILED DESCRIPTION:
Decades of immunosuppressive drug development has produced an array of powerful pharmacological agents, but the various drawbacks associated with these treatments leaves considerable room for improvement. By harnessing the power of suppressive mechanisms in the human immune system, regulatory cell therapy may be able to support peripheral tolerance and induce a level of donor-specific unresponsiveness that allows for a reduction in the use of conventional immunosuppression in organ transplant recipients. Several alternative regulatory cell types have been identified as potential adjunct immunotherapies for solid organ transplantation and are now approaching a stage of development that would allow clinical testing in an early-stage trial. The EU-funded international ONE Study consortium aims to answer the question as to whether M reg treatment, or other immunoregulatory cell-based therapies, can be advanced in the clinical management of solid organ transplant recipients.

This particular M reg trial aims to explore the potential of M reg therapy as an adjunct immunosuppressive treatment in living-donor renal transplant recipients through a clinical protocol design shared by other investigators in The ONE Study group testing additional regulatory cell therapies in separate trials.

ELIGIBILITY:
RECIPEINT

Inclusion Criteria:

* Chronic renal insufficiency necessitating kidney Tx
* Aged at least 18 years
* Able to commence the immunosuppressive regimen as specified
* Willing and able to participate in The ONE Study subprojects
* Signed and dated written informed consent

Exclusion Criteria:

* Patient has previously received any tissue or organ Tx
* Known contraindication to the protocol-specified treatments /medications
* HLA 0-0-0 mismatch
* PRA grade >40% within 6 mo. prior to enrolment
* Previous desensitisation treatment
* Concomitant malignancy or history of malignancy <5 years before study entry (excluding successfully-treated non-metastatic skin BCC or SCC)
* Significant local or systemic infection
* HIV-positive, EBV-negative or suffering chronic viral hepatitis
* CMV negative and receiving a kidney from a CMV+ donor
* Significant liver disease
* Malignant or pre-malignant haematological conditions
* Any uncontrolled condition that could interfere with study objectives
* Any condition placing the subject at undue risk
* Ongoing treatment with systemic immunosuppressive drugs at study entry
* Exposure to an investigational product during the study, or within 28 days or 5 half-lives of the product before study entry
* Female patients of child-bearing potential with a +pregnancy test
* Female patients breast-feeding or that are of child bearing potential and unwilling to use effective birth control
* Psychological, familial, sociological or geographical factors hampering compliance
* Any substance abuse or psychiatric disorder
* Patients unable to freely give informed consent
* Known IgA or IgG deficiency
* Any pro-coagulant disposition causing undue risk
* Previous history of transfusion-associated disease causing undue risk
* Conditions resulting in substantially reduced pulmonary vasculature or increased pulmonary vascular resistance. Diseases causing substantially elevated pulmonary arterial or right heart hypertrophy or dysfunction
* Known atrial or ventricular septal defects posing a risk of embolism
* Known hypersensitivity to components of the manufactured cell product

DONOR

Inclusion Criteria:

* Eligible for live kidney donation
* Aged at least 18 years
* Willing and able to provide a blood sample for The ONE Study Subproject
* Willing to provide personal and medical/biological data for the trial analysis
* Eligible for leucapheresis prior to organ donation
* Signed and dated written informed consent

Exclusion Criteria:

* Genetically identical to the prospective organ recipient at the HLA loci (0-0-0 mismatch)
* CMV-positive and donating to a CMV-negative recipient
* Exposure to an investigational product during the study, or within 28 days or 5 half-lives of the product before study entry
* Any form of substance abuse, psychiatric disorder, or other condition that, in the opinion of the Investigator, may invalidate communication with the investigator and/or designated study personnel
* Subjects unable to freely give their informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2014-07-24 (Actual); Primary Completion 2018-12-03 (Actual); Study Completion 2018-12-03 (Actual)

PRIMARY OUTCOMES:
biopsy-confirmed acute rejection incidence | 60 weeks

SECONDARY OUTCOMES:
time to first acute rejection episode | 60 weeks
severity of acute rejection episodes | 60 weeks
  based on response to treatment and histological scoring
total immunosuppressive burden | 60 weeks
  assessed at last study visit
incidence of patients treated for subclinical acute rejection | 60 weeks
prevention of chronic graft dysfunction (chronic rejection or IF/TA) | 60 weeks
  assessed by clinical (impairment of GFR) and histopathological (Banff staging) measures
incidence of post-transplant dialysis, inclusion on the transplant waiting list or re-transplantation following graft loss through rejection | 60 weeks
avoidance of drug-related complications by immunosuppressant reduction | 60 weeks
  assessed by the incidence of reported adverse drug reactions
incidence of embolic pulmonary complications and other embolic events | 60 weeks
incidence of immunological reactions resulting in anaphylactoid reactions, immediate cardiovascular compromise or other acute organ failure | 1 week
biochemical disturbances caused by cell infusion | 1 week
over-suppression of the immune system assessed by the incidence of major and/or opportunistic infections, especially CMV, EBV and polyoma virus | 60 weeks
over-suppression of the immune system assessed by the incidence of neoplasia | 60 weeks
immunological condition of study patients | 60 weeks
  an extensive immune monitoring program has been established in The ONE Study

OTHER OUTCOMES:
incidence of malignancies arising directly from Mreg_UKR | 60 weeks
incidence of autoimmune disorders | 60 weeks
incidence of inflammatory pathologies | 60 weeks
incidence of anaemia, cytopaenia or biochemical disturbances unrelated to the function of the transplanted kidney | 60 weeks
A Health-Economics Subproject will evaluate the health-related quality-of-life of trial patients using patient-reported outcome measures | 60 weeks
  this subproject will also calculate the cost-effectiveness of the Mreg_UKR cell product

CONTACTS AND LOCATIONS:
Overall Officials: Edward K Geissler, PhD, Study Director — University Hospital Regensburg, University of Regensburg; Bernhard Banas, MD, Principal Investigator — University Hospital Regensburg, University of Regensburg; James A Hutchinson, MD, PhD, Principal Investigator — University Hospital Regensburg, University of Regensburg
Locations (1):
- University Hospital Regensburg, Regensburg, Germany

REFERENCES:
- [Background] Geissler EK. The ONE Study compares cell therapy products in organ transplantation: introduction to a review series on suppressive monocyte-derived cells. Transplant Res. 2012 Sep 28;1(1):11. doi: 10.1186/2047-1440-1-11. No abstract available. PMID 23369457
- [Derived] Sawitzki B, Harden PN, Reinke P, Moreau A, Hutchinson JA, Game DS, Tang Q, Guinan EC, Battaglia M, Burlingham WJ, Roberts ISD, Streitz M, Josien R, Boger CA, Scotta C, Markmann JF, Hester JL, Juerchott K, Braudeau C, James B, Contreras-Ruiz L, van der Net JB, Bergler T, Caldara R, Petchey W, Edinger M, Dupas N, Kapinsky M, Mutzbauer I, Otto NM, Ollinger R, Hernandez-Fuentes MP, Issa F, Ahrens N, Meyenberg C, Karitzky S, Kunzendorf U, Knechtle SJ, Grinyo J, Morris PJ, Brent L, Bushell A, Turka LA, Bluestone JA, Lechler RI, Schlitt HJ, Cuturi MC, Schlickeiser S, Friend PJ, Miloud T, Scheffold A, Secchi A, Crisalli K, Kang SM, Hilton R, Banas B, Blancho G, Volk HD, Lombardi G, Wood KJ, Geissler EK. Regulatory cell therapy in kidney transplantation (The ONE Study): a harmonised design and analysis of seven non-randomised, single-arm, phase 1/2A trials. Lancet. 2020 May 23;395(10237):1627-1639. doi: 10.1016/S0140-6736(20)30167-7. PMID 32446407
- See also: ONE Study — http://www.onestudy.org